CLINICAL TRIAL: NCT05634655
Title: Dissecting the Mechanism of DNA Methylation on the Invasiveness of Pituitary
Brief Title: Dissecting the Mechanism of DNA Methylation on the Invasiveness of Pituitary Tumors.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0765
Record Dates: First submitted 2022-11-23; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2021-12

CONDITIONS: Pituitary Tumors
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — tissues of pititary adenomas
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- invasive PAs
  Interventions: Other: no interventions between two groups
- non-invasive PAs
  Interventions: Other: no interventions between two groups

INTERVENTIONS:
Other: no interventions between two groups — no interventions between two groups

SUMMARY:
DNA methylation is one of the important ways of protein post-translational modification.Pituitary adenoma (PA) is a benign neuroendocrine tumor that originates from adenohypophysial 45 cells, and accounts for 10%-20% of all primary intracranial tumors. However some PAs can present with high invasiveness and irregular growth, which tend to compresses the optic chiasm and third ventricle, encase the internal carotid artery, and affect hormone secretion from the pituitary gland and hypothalamus. In this study we focus on the mechanism of DNA methylation on the invasiveness of pituitary tumors.

ELIGIBILITY:
Inclusion Criteria:

* 1) histologically confirmed PAs, 2) Non-function pituitary adenomas

Exclusion Criteria:

* 1) Associated with other tumors or serious underlying diseases, 2) the medical records were not complete, or the follow-up data were missing.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients with PAs who underwent TSS at The Second Affiliated 62 Hospital Zhejiang University School of Medicine was retrospectively analyzed.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Residual tumor size | 1 week after surgery
  Tumor size was evaluated by postoperative MRI
tumor recurrence | three years
  During the follow-up, the tumor recurrence was observed closely

CONTACTS AND LOCATIONS:
Locations (1):
- 2ndAffiliated Hospital, School of Medicine, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No